CLINICAL TRIAL: NCT00337181
Title: Extended Evaluation of the Virologic, Immunologic, and Clinical Course of Volunteers Who Become HIV-1 Infected During Participation in a Phase III Vaccine Trial of ALVAC-HIV and AIDSVAX® B/E.
Brief Title: Follow up of Thai Adult Volunteers With Breakthrough HIV Infection After Participation in a Preventive HIV Vaccine Trial
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Royal Thai Ministry of Public Health (Unknown); Mahidol University (Other); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: A-11048; RV152 (Other: WRAIR)
Record Dates: First submitted 2006-06-14; First posted 2006-06-15 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: HIV-1
Keywords: HIV-1; Natural History; HIV vaccine; Thailand

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccine Group: Received vaccination in RV144
- Placebo Group: Received placebo in RV144

SUMMARY:
This protocol will study the clinical course of HIV-infection among volunteers who have received either a placebo injection or the experimental vaccine combination of ALVAC-HIV and AIDSVAX B/E prior to HIV-1 infection in reference to study NCT00223080 RV144. The study will assess whether those who received the experimental vaccine combination have a slower progression of HIV disease compared to those who received the placebo injection.

DETAILED DESCRIPTION:
Prospective cohort study of the clinical course of HIV-1 infection occurring after candidate HIV-1 vaccination (breakthrough infection) with ALVAC-HIV (vcP1521) and AIDSVAX B/E in reference to study NCT00223080 RV144. This study will enroll volunteers who become HIV-infected during the course of follow up in a phase III preventive HIV vaccine trial conducted in Rayong and Chon Buri, Thailand. Volunteers will be enrolled in this protocol to provide additional long-term follow up to establish whether differences in viral load after infection (comparing vaccine to placebo) are associated with altered disease outcomes, as well as provide more detailed immunologic and virologic assessment of these volunteers.

After enrollment in RV152, follow-up visits were scheduled at 0, 1, 3, and 6 months, and every 3 months thereafter. After month 12, CD4+ T cell counts and viral load were obtained at 6-month intervals until the CD4+ T cell count declined to <350/ul or highly-active antiretroviral therapy (HAART) was initiated, at which time CD4+ T cell counts and viral load were obtained every 3 months. Peripartum antiretroviral drugs given for prevention of mother-to-child-transmission was not considered a study endpoint, however HAART initiated during pregnancy and continued post-partum was counted. After a single CD4+ T-cell count < 350/ul a second sample was requested about 2 weeks later, and if the confirmatory measurement was >350/ul, a study endpoint was not registered and the volunteer resumed a normal visit schedule. A single genital fluid collection for viral load was obtained at the first RV152 visit. Clinical and laboratory data from RV144, including CD4+ T-cell and HIV-1 plasma viral load measurements, were linked to RV152 to inform primary and secondary protocol analyses as well as volunteer care and treatment.

ELIGIBILITY:
Inclusion Criteria:

* All individuals who become HIV-infected after receiving experimental vaccine or placebo in the RV144 clinical trial if they received at least one injection.
* The volunteer must give written, informed consent.

Exclusion Criteria:

* Persons who have a medical or psychiatric disorder, that in the judgment of the investigator(s), would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent.
* Persons who become HIV-infected after the completion of the RV144 protocol.

Ages: 18 Years to 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All individuals who became HIV-infected after receiving experimental vaccine or placebo in the RV144 clinical trial if they received at least one injection
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Supachai Rerks-Ngarm, MD, Principal Investigator — Ministry of Health, Thailand
Locations (1):
- Chon Buri Regional Hospital, Chon Buri, Chon Buri Province, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rerks-Ngarm S, Paris RM, Chunsutthiwat S, Premsri N, Namwat C, Bowonwatanuwong C, Li SS, Kaewkungkal J, Trichavaroj R, Churikanont N, de Souza MS, Andrews C, Francis D, Adams E, Flores J, Gurunathan S, Tartaglia J, O'Connell RJ, Eamsila C, Nitayaphan S, Ngauy V, Thongcharoen P, Kunasol P, Michael NL, Robb ML, Gilbert PB, Kim JH. Extended evaluation of the virologic, immunologic, and clinical course of volunteers who acquired HIV-1 infection in a phase III vaccine trial of ALVAC-HIV and AIDSVAX B/E. J Infect Dis. 2013 Apr 15;207(8):1195-205. doi: 10.1093/infdis/jis478. Epub 2012 Jul 26. PMID 22837492

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccine Group | Placebo Group
Started | 49 | 65
Completed | 49 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 49 | 65 | 114
Age, Customized [Count of Participants; unit: Participants]
  <20 | 12 | 10 | 22
  21-25 | 18 | 33 | 51
  >26 | 19 | 22 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 28 | 47
  Male | 30 | 37 | 67
Region of Enrollment [Number; unit: participants]
  Thailand | 49 | 65 | 114
Calendar year of infection diagnosis [Count of Participants; unit: Participants]
  2004-2005 | 13 | 17 | 30
  2006 | 13 | 26 | 39
  2007 | 17 | 10 | 27
  2008-2009 | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching Clinical Long Term Component Endpoints
Description: Evaluate the vaccine effect on clinical long term endpoints: CD4 is for CD4<350 endpoint; ART is for initiation of highly-active antiretroviral therapy (HAART) endpoint; ADI is for AIDS-defining illness endpoint; A combination of multiple endpoints is listed in order of occurrences of the endpoints
Time Frame: 66 months
Population: Participants analyzed correlates to responders of endpoints
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine Group | Placebo Group
Number analyzed (Participants) | 26 | 35
Participants
  CD4 <350 only (CD4) | 3 | 5
  CD4-ART | 18 | 23
  CD4-ADI | 0 | 0
  CD4-ART-ADI | 1 | 1
  CD4-ADI-ART | 1 | 2
  ART Initiation only (ART) | 1 | 3
  ART-CD4 | 1 | 0
  ART-ADI | 0 | 0
  ART-CD4-ADI | 0 | 0
  ART-ADI-CD4 | 0 | 0
  AIDS Illness only (ADI) | 0 | 0
  ADI-CD4 | 0 | 0
  ADI-ART | 0 | 0
  ADI-CD4-ART | 1 | 1
  ADI-ART-CD4 | 0 | 0

ADVERSE EVENTS:
Description: A final report can't be located for this protocol. Results info was pulled from an abstract published after study completion. AEs were not referenced in the abstract so therefore there are no AEs to report.
Arm/Group | Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
A final report can't be located for this protocol. Results were pulled from an abstract that was published after completion. Outcome endpoints in protocol description will not match final outcome measures in results section. AE's can't be located.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No